CLINICAL TRIAL: NCT04962802
Title: Evaluation of Manhood 2.0: A Community-Based Teen Pregnancy Prevention Program for Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: Promundo, United States (Other); Latin American Youth Center (Unknown)
Responsible Party: Principal Investigator, Jennifer Manlove, Senior Program Area Director, Child Trends
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5U01DP006129 (NIH)
Record Dates: First submitted 2021-07-10; First posted 2021-07-15 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Sexual Behavior; Unprotected Sex
MeSH Terms: conditions — Sexual Behavior; Unsafe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manhood 2.0 (Experimental): Manhood 2.0 is a group-level intervention, delivered in 7 sessions over 13 hours, and is based on social cognitive theory, social norm theory, theory of gender and power, and the theory of reasoned action. Sessions were delivered twice a week, for approximately 3.5 weeks. For the final session, participants received one hour of content and were administered the immediate post-intervention survey. The intervention takes a holistic, gender-transformative approach, includes reproductive health knowledge, healthy relationships, altering gender norms and stereotypes which drive reproductive health behavior, and explicit and proactive support of female partner contraceptive use. Activities are designed to engage young men in critical reflection and dialogue about gender norms, and then apply these discussions to a range of key issues including intimate relationships, gender-based violence, substance abuse, STIs, and early pregnancy.
  Interventions: Behavioral: Manhood 2.0
- Post-High School Readiness (Placebo Comparator): The Post-High School Readiness Program helped youth build skills around identifying colleges or programs of interest, completing applications for programs, writing resumes and increasing financial literacy. The post-high school readiness curriculum was delivered by LAYC staff members and the content was delivered twice a week, for approximately 3.5 weeks (as with the intervention). For the final session, participants did not receive content and were administered the immediate post-intervention survey.
  Interventions: Behavioral: Post-High School Readiness

INTERVENTIONS:
Behavioral: Manhood 2.0 — Manhood 2.0 engages young men in questioning, challenging, and transforming harmful gender norms, with the goal of reducing intimate partner and sexual violence and unintended teen pregnancy. Manhood 2.0 is a male-only group-level intervention, based on social cognitive theory, social norm theory, theory of gender and power, and the theory of reasoned action. Activities include group discussion, role playing, knowledge sharing, and skill-building; their purpose is to challenge young men to think critically about social expectations and restrictive norms, engage in dialogue about these gender norms, and then assess the way rigid norms affect their attitudes and behaviors toward key issues, including intimate relationships, gender-based violence, substance abuse, sexually transmitted infections, and early pregnancy. Sessions are two hours long and occur once a week for seven weeks.
  Arms: Manhood 2.0
Behavioral: Post-High School Readiness — Post-High School Readiness program helps young men prepare for life after high school. This includes helping them prepare resumes, learning how to apply to jobs or colleges, providing interview prep, and other life skills. It is a male-only group-level program that includes discussion, feedback, knowledge sharing, and skill-building; their purpose is to prepare young men for life after high school. Sessions are two hours long and occur once a week for seven weeks.
  Arms: Post-High School Readiness

SUMMARY:
Manhood 2.0 is a male-only group-level intervention, delivered over 13 hours, based on social cognitive theory, social norm theory, theory of gender and power, and the theory of reasoned action. The intervention is a gender-transformative program that promotes critical reflection and awareness on reproductive health, healthy relationships, gender norms and stereotypes that drive reproductive health behavior, and explicit and proactive support of female partner contraceptive use. Activities include group discussion, role playing, knowledge sharing, and skill-building; their purpose is to challenge young men to think critically about social expectations and restrictive norms, engage in dialogue about these gender norms, and then assess the way rigid norms affect their attitudes and behaviors toward a number of key issues, including intimate relationships, gender-based violence, substance abuse, sexually transmitted infections, and early pregnancy. Young men receive the intervention at a local community center or high school. Comparison condition young men receive a post-high school readiness program that does not discuss gender norms or sexual and reproductive health. The study was conducted with six cohorts of eligible young men ages 15-18 who received a baseline, immediate post-intervention, and three-month post-intervention survey. To participate in the study, individuals had to meet all the following criteria: (1) Identify as male; (2) Ages 15 to 18; (3) Not actively planning a pregnancy with someone; (4) Never participated in the community center's sexual and reproductive health program; (5) Received no additional sexual or reproductive health programming in the last three months; (6) Able to participate in a program delivered in English only.

The investigators hypothesized that Manhood 2.0 participants would have lower rates of unprotected sex and more equitable attitudes towards gender than comparison participants.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages 15-18
* Able to participate in a program delivered only in English

Exclusion Criteria:

* Actively planning a pregnancy with someone
* Received sexual and reproductive health programming in the last 3 months
* Ever participated in the intervention site's sexual and reproductive health program

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Unprotected sex | 1.5 months after baseline
  Number of participants who reporting having vaginal sex in the past month without using a condom or other contraceptive method.
Unprotected sex | 4.5 months after baseline
  Number of participants who reporting having vaginal sex in the past month without using a condom or other contraceptive method.
Sex without a condom | 1.5 months after baseline
  Number of participants who reporting having vaginal sex in the past month without using a condom.
Sex without a condom | 4.5 months after baseline
  Number of participants who reporting having vaginal sex in the past month without using a condom.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Manlove, PhD, Principal Investigator — Child Trends
Locations (1):
- Latin American Youth Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No